CLINICAL TRIAL: NCT03649100
Title: Does the New Hydrophilic Surface Have Any Influence on Early Success Rate and Implant Stability During Osseointegration Period? A Split-mouth, Randomised Controlled Trial
Brief Title: Osseointegration With a New Hydrophilic Surface
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osstem AIC (Other)
Responsible Party: Principal Investigator, Marco Tallarico, Principal investigator, Osstem AIC
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Osstem_002
Record Dates: First submitted 2018-08-17; First posted 2018-08-28 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Dental Implant Stability
Keywords: Dental implants; Implant stability; Osseointegration; ISQ measurement

STUDY DESIGN:
Intervention Model Description: To randomly compare implant stability quotient (ISQ) of Hiossen ET III implants with its new hydrophilic surface (NH) and Hiossen ET III implants with the conventional SA surface, in a split-mouth randomized study.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: A blinded collaborator opened the opaque envelope after implant site development, giving the implant to the investigator that remain blinded. Both the test and control implants are perfectly the same.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hiossen ET III NH implant (Experimental): Implant placement, dental implant with Sandblasted and Acid-etched (SA) surface implant and newly developed bio-absorbable apatite nano coating (Hiossen ET III NH implant, NH group)
  Interventions: Procedure: Implant placement
- Hiossen ET III SA implant (Active Comparator): Implant placement, dental implant with the conventional sandblasted and Acid-etched (SA) surface implant (Hiossen ET III Sto arrivando! implant, Sto arrivando! group)
  Interventions: Procedure: Implant placement

INTERVENTIONS:
Procedure: Implant placement — Conventional implant placement. Implant site development was prepared according to the manufacturer's instruction by the investigator, before knowing the randomized implant (NH or SA).

SUMMARY:
This study was conducted to compare implant stability of Hiossen ET III implants with its new hydrophilic surface (NH) and Hiossen ET III implants with the SA surface.

DETAILED DESCRIPTION:
Patients required at least two teeth to be rehabilitated with a fixed, implant-supported restoration, consecutively enrolled. Patients randomly received Sandblasted and Acid-etched (SA) surface implants (SA group) or SA implants with a newly developed bio-absorbable apatite nano coating (NH group). Outcome measures were: implant and prosthetic survival rate, complications, insertion torque, and implant stability quotient (ISQ) measured at implant placement and every week up to 8 weeks after implant placement. Comparison between groups was made by unpaired t test, while comparison between each follow-up will be made by paired t tests to detect any change during the follow-up. Complications and failures were compared by using Fisher exact test.

ELIGIBILITY:
Inclusion Criteria:

* Any healthy patients
* Aged 18 years or older
* Requiring at least two implants to be rehabilitated with a fixed implant supported restoration
* Full mouth bleeding and full mouth plaque index lower than or equal to 25%
* Sufficient bone to allow placement of at least 11.5 mm-long implants, and bone width of at least six to eight mm for the placement of a regular platform Hiossen ET III implant (Deutsche Osstem GmbH, Eschborn, Germany).

Exclusion Criteria:

* Positive medical findings
* Psychiatric therapy
* Pregnancy or nursing
* Smoking more than 10 cigarettes per day
* Insertion torque < 35 Ncm
* Untreated periodontitis
* Acute and chronic infections of the adjacent tissues or natural dentition
* Previous radiotherapy of the oral and maxillofacial region within the last five years
* Post-extractive implants (at least three months after tooth extraction)
* Absence of teeth in the opposing jaw
* Severe clenching or bruxism
* Severe maxillo-mandibular skeletal discrepancy
* Poor oral hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Implant and prosthetic success rates | 4 months after implant placement (baseline)
  Success rates of the implants and prostheses were evaluated by an independent assessor (EX). An implant was considered a failure if it presented mobility, assessed after the osseointegration period by tapping or rocking the implant head with the metallic handles of two instruments, progressive marginal bone loss or infection, or any mechanical complications rendering the implant unusable, although still mechanically stable in the bone. A prosthesis was considered a failure if it needed to be replaced with another prosthesis.

SECONDARY OUTCOMES:
Technical or biological complications | 4 months after implant placement
  Any biological complication, such as pain, swelling, and or suppuration, as well as any technical complication, such as screw loosening, fracture of the framework and/or the veneering material will be recorded during the follow-up period. Complications were evaluated and treated by the same surgeon (MT).
Implant stability quotient (ISQ) | Each week (after implant placement) up to 8 weeks, and then 12 weeks (after implant placement)
  Implant stability quotient (ISQ) values were recorded each week up to 8 weeks, and then after 12 weeks, using resonance frequency analysis (Osstell Mentor device, Osstell, Gothenburg, Sweden). Each implant was measured twice. First in a messy-distal direction and then in a buck-lingual direction. The mean value was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tallarico, Dr, Principal Investigator — Osstem AIC
Locations (3):
- Italy (3):
  - Nicola Baldini, Florence
  - Fulvio Gatti, Milan
  - Studio Odontoiatrico Marco Tallarico, Rome

IPD SHARING:
Plan to Share IPD: No